CLINICAL TRIAL: NCT05640167
Title: EMPOWER PD - Feasibility of an Interdisciplinary Clinic for People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Collaborators: Brown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1929810-1
Record Dates: First submitted 2022-11-18; First posted 2022-12-07 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: Patient-centric care; Interdisciplinary care; Parkinson Disease education
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EMPOWER PD Clinic Participation (Other): All participants will be assigned to the same interdisciplinary clinic and educational intervention
  Interventions: Behavioral: Interdisciplinary Clinic

INTERVENTIONS:
Behavioral: Interdisciplinary Clinic — Interdisciplinary Clinic - assessment and recommendations by Nutrition, Pharmacy, Physical Therapy, and Speech Therapy and Educational Seminar - Parkinson's specific education and resources in group format

SUMMARY:
This study is a nonrandomized, pilot study of an interdisciplinary, patient-centric model of health care delivery in a "boot camp" style structured clinic for people diagnosed with Parkinson's disease (PwPD). 20 participants will attend a three session EMPOWER PD clinic and a two month follow up interview. The primary objective is to assess feasibility and acceptability of the newly developed clinic intervention as well as individual perception of experience and barriers.

DETAILED DESCRIPTION:
This study is a nonrandomized, pilot study of an interdisciplinary, patient-centric model of health care delivery in a "boot camp" style structured clinic for people diagnosed with Parkinson's disease (PwPD). 20 participants will attend a three session EMPOWER PD clinic and a two month follow up interview.

Participants will receive a comprehensive assessment by each member of an interdisciplinary team including physical therapy, speech therapy, nutrition, social work or psychology, and pharmacy. Participants will return the following week for a half day educational symposium. This is a group format and they will receive a session from each of the disciplines covering topics such as exercise, nutrition, communication, socialization, sleep hygiene, medication management, and coping. The final clinic session will be a one hour 1:1 meeting where individualized recommendations will be provided. A participant identified caregiver is invited/allowed to accompany the participant throughout the assessment and educational process whenever possible however, no information or questionnaires are being collected from them.

The primary objective is to assess feasibility and acceptability of the newly developed clinic intervention as well as individual perception of experience and barriers with data derived from a program survey and semi-structured interview completed two months after clinic completion. Secondary objectives will test patient response to clinic intervention related to self-reported outcome measures (SROs) including Patient Centered Outcome Questionnaire PD, PD Knowledge, quality of life, fatigue, confidence with balance, and self-efficacy for exercise.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of idiopathic Parkinson Disease
* Living in the community (not institutionalized)

Exclusion Criteria:

* A diagnosis of atypical Parkinsonism
* Institutionalized (living in a nursing home setting)

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Clarkin, PhD, Principal Investigator — University of Rhode Island
Locations (1):
- University of Rhode Island - Physical Therapy Department, Kingston, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-three individuals were screened for the clinic. Two were unable to attend due to limited weekend availability of the clinic, a third could not attend due to geographic/driving barriers, and the remaining 20 were confirmed to attend the EMPOWER PD Clinic in one of two locations offered. One individual was a no show to the clinic resulting in 19 participants enrolled in the study.
Groups:
- EMPOWER PD Clinic Participation: All participants were assigned to the same interdisciplinary clinic and educational intervention.
  Interdisciplinary Clinic: Interdisciplinary Clinic - assessment and recommendations by Nutrition, Pharmacy, Physical Therapy, and Speech Therapy and Educational Seminar - Parkinson's specific education and resources in group format
Period: Overall Study
Arm/Group | EMPOWER PD Clinic Participation
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- EMPOWER PD Clinic Participation: All participants were assigned to the same interdisciplinary clinic and educational intervention
  Interdisciplinary Clinic: Interdisciplinary Clinic - assessment and recommendations by Nutrition, Pharmacy, Physical Therapy, and Speech Therapy and Educational Seminar - Parkinson's specific education and resources in group format
Arm/Group | EMPOWER PD Clinic Participation
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.53 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19
Education level [Count of Participants; unit: Participants]
  Up to High School or GED | 2
  Some College or Vocational School | 5
  College degree | 12
Years Living with Parkinson's Disease [Mean (Standard Deviation); unit: years] — This is the number of years an individual had been living with Parkinson's disease based on the year they were diagnosed by a physician. This self reported by the participant and collected during the intake process.
  years | 6.1 (5.45)
Stage of Parkinson's Disease [Count of Participants; unit: Participants] — The number of years living with Parkinson's disease was used to categorize what stage of the disease an individual was in. Early stage was defined as 0-4 years, mid stage was 5-10 years, and advanced was greater than 10 years.
  Participants
    Early Stage (0-4 years) | 9
    Mid Stage (5-10 years) | 6
    Adavanced Stage (>10 years) | 4
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) is a cognitive screen to assess baseline cognitive level across several domains. MOCA scale is scored from 0 (lowest cognitive functioning) to 28 (highest cognitive functioning) with a cut off score of <26 to detect Mild cognitive impairment. This was collected during the interdisciplinary clinic component.
  units on a scale | 26.26 (4.98)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Accessibility
Description: Feasibility is measured by attendance and retention and survey completion rates. Attendance reported for each component of the clinic (clinic, seminar, 1:1 meeting, and follow-up interview). Retention reflects the number of participants that participated in all 4 components. Survey completion rates reflect the number of participants that completed all self report measures at Baseline and End of Study.
Time Frame: Baseline and End of Study - 2 Months
Measure: Count of Participants; unit: Participants
Arm/Group | EMPOWER PD Clinic Participation
Number analyzed (Participants) | 19
Participants
  Attendance Clinic | 19
  Attendance Seminar | 19
  Attendance 1:1 | 19
  Attendance Interview | 19
  Retention Rate | 19
  Survey Completion Baseline | 18
  Survey Completion End of study | 18

2. Primary Outcome: Feasibility: Program Survey
Description: A series of 12 statements regarding acceptability, process, barriers, and perception of experience of clinic will be scored by participants on a scale of 1 (disagree) to 5 (agree) with a higher score on each statement indicating more positive outcome. The average response per question is reported below.
Time Frame: End of Study - 2 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EMPOWER PD Clinic Participation
Number analyzed (Participants) | 19
units on a scale
  Question 1 - The clinic was located in an area of RI that was accessible to me. | 4.947 (0.229)
  Question 2 - Parking was easy and accessible | 4.947 (0.229)
  Question 3 - The building where I attended the clinic was accessible. | 4.947 (0.229)
  Question 4 - The clinic was well organized. | 4.947 (0.229)
  Question 5 - It was helpful to be seen by the physical therapist. | 4.947 (0.229)
  Question 6 - It was helpful to be seen by the speech language pathologist. | 4.894 (0.315)
  Question 7 - It was helpful to be seen by the nutritionist. | 4.842 (0.501)
  Question 8 - It was helpful to be seen by the pharmacist. | 4.789 (0.535)
  Question 9 - The four-hour educational seminar increased my knowledge | 4.789 (0.418)
  Question 10 - I feel more confident with my ability to access resources in RI | 4.578 (0.60)
  Question 11 - I have made progress on the individual goals I identified during the clinic | 4.368 (0.683)
  Question 12 - Participating in EMPOWER PD added value to my ability to manage my Parkinson's disease | 4.842 (0.374)

3. Primary Outcome: Change in Patient Centered Outcome Questionnaire
Description: Parkinson's Disease (PCOQ-PD) The PCOQ-PD evaluates treatment success and expectations from the patient's perspective across 10 motor and non-motor functional domains grouped into four sections. Patients are asked to rate for each domain with each section: (1) their usual levels of self-defined difficulty over the past week, (2) their success criteria for treatment outcomes, (3) their expectations for their treatment, regardless of their previous treatment experiences, and (4) how important it was for them to see improvement. Participants used a 101-point numerical rating scale to indicate their rating, anchored by 0 ("None") to 100 ("Worst Imaginable") for the first three sections and by 0 ("Not at All Important") to 100 ("Most Important") for the fourth section. The mean response and standard deviation are reported below.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMPOWER PD Clinic Participation
Number analyzed (Participants) | 19
score on a scale
  Pain - Importance | 34.47 (9.22)
  Fatigue - Importance | 50.26 (8.25)
  Emotional Distress - Importance Emotional Distress - Importance | 33.16 (8.21)
  Interference with ADLs - Importance | 41.48 (8.17)
  Tremor - Importance | 36.58 (7.99)
  Stiffness - Importance | 56.05 (8.72)
  Slowness - Importance | 45.53 (8.39)
  Walking Problems - Importance | 51.32 (9.23)
  Thnking Porblems - Importance | 51.84 (9.15)
  Sleep Problems - Importance | 38.95 (8.57)

4. Primary Outcome: Parkinson's Disease Knowledge Questionnaire
Description: Knowledge regarding Parkinson's disease as measured by the Parkinson's Disease Knowledge Questionnaire (PDKQ). Participants indicate their knowledge of 26 items related to Parkinson's disease with a true or false response.
Time Frame: Baseline and End of Study - 2 months
Population: One participant was dropped from the analysis due to cognitive impairment and difficulty completing the questionnaire
Measure: Mean (Standard Deviation); unit: percentage of correct answers
Arm/Group | EMPOWER PD Clinic Participation
Number analyzed (Participants) | 18
percentage of correct answers
  PDKQ Pre-Assess | 66.03 (10.23)
  PDKQ Post-Assess | 75.21 (12.32)
Statistical Analysis 1: Comparison: EMPOWER PD Clinic Participation; Test type: Other; p = 0.015, t-test, 2 sided; Degrees of freedom 17

5. Primary Outcome: Change in Health Education Impact Questionnaire
Description: Subjects score 42 items across 8 domains using a Likert-style question format indicated their strength of agreement by checking an option from 1 ("strongly disagree") through 5 ("strongly agree").
Time Frame: Baseline and End of Study - 2 Months
Population: One participant was dropped from the analysis due to cognitive impairment and difficulty completing the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale 1 to 5
Arm/Group | EMPOWER PD Clinic Participation
Number analyzed (Participants) | 18
score on a scale 1 to 5
  Postive engagement - Pre Assess | 3.78 (.85)
  Postive engagement - Post Assess | 4.18 (.73)
  Health directed activities - Pre Assess | 3.28 (.4)
  Health directed activities - Post Assess | 3.58 (.42)
  Skill and Technique Aquisition - Pre Assess | 3.02 (.21)
  Skill and Technique Aquisition - Post Assess | 3.32 (.39)
  Constructive Attitudes - Pre Assess | 3.22 (.38)
  Constructive Attitudes - Post Assess | 3.67 (.34)
  Self monitoring and insight - Pre Assess | 3.13 (.20)
  Self monitoring and insight - Post Assess | 3.48 (.35)
  Health service navigation - Pre Assess | 3.22 (.34)
  Health service navigation - Post Assess | 3.47 (.55)
  Social integration and support - Pre Assess | 3.14 (.35)
  Social integration and support - Post Assess | 3.37 (.55)
  Emotional well-being - Pre Assess | 2.93 (.25)
  Emotional well-being - Post Assess | 2.70 (.52)
Statistical Analysis 1: Comparison: EMPOWER PD Clinic Participation; Test type: Other; p = 0.114, t-test, 2 sided — Positive p = 0.114 Health-directed p = 0.028 Skill and Technique p = 0.013 Constructive attitudes p = 0.003 Self-monitoring & insight p = 0.001 Health service navigation p = 0.077 Social Integration p = 0.126 Emotional well-being p = 0.093

6. Secondary Outcome: Change in Self-Efficacy for Exercise
Description: Self-Efficacy for Exercise scale consists of nine situations (weather, boredom, exercising alone, not pleasurable, too busy, feel tired, stress, depressed) that might effect participation in exercise For each situation, the subject uses the scale from 0 (not confident) to 10 (very confident) to describe their current confidence that they could exercise 3 times a week for 20 minutes each time. Total score is calculated by summing the responses to each question. This scale has a range of total scores from 0-90. A higher score indicates higher self-efficacy for exercise. Participants total score was then divided by 90 to convert to a percentage.
Time Frame: Baseline and End of Study - 2 Months
Population: One participant was dropped from the analysis due to cognitive impairment and difficulty completing the questionnaire
Measure: Mean (Standard Deviation); unit: percentage of agreement with statements
Arm/Group | EMPOWER PD Clinic Participation
Number analyzed (Participants) | 18
percentage of agreement with statements
  Self-Efficacy for Exercise - Pre Assess | 64.82 (20.77)
  Self-Efficacy for Exercise - Post Assess | 67.10 (20.88)
Statistical Analysis 1: Comparison: EMPOWER PD Clinic Participation; Test type: Other; p = 0.59, t-test, 2 sided

7. Secondary Outcome: Change in Balance Confidence Measured With the Activities-specific Balance Confidence (ABC) Scale.
Description: The ABC is The ABC is an 16 question survey and ratings should consist of whole numbers (0-100) for each item. Total the ratings (possible range = 0 - 1600) and divide by 16 to get each subject's ABC score which is a percentage of agreement out of 100%.
Time Frame: Baseline and End of Study - 2 Months
Population: One participant was dropped from the analysis due to cognitive impairment and difficulty completing the questionnaire
Measure: Mean (Standard Deviation); unit: percentage of agreement with statements
Arm/Group | EMPOWER PD Clinic Participation
Number analyzed (Participants) | 18
percentage of agreement with statements
  ABC Pre Assess | 80.79 (15.41)
  ABC Post Assess | 85.37 (12.74)
Statistical Analysis 1: Comparison: EMPOWER PD Clinic Participation; Test type: Other; p = 0.03, t-test, 2 sided

8. Secondary Outcome: Change in Quality of Life Measured With the Parkinson Disease Questionnaire-39 (PDQ-39)
Description: The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month covering 8 dimensions scored on a 5 point ordinal system (0=never, 4=always). Dimension score = sum of scores of each item in the dimension divided by the maximum possible score of all the items in the dimension, multiplied by 100. Each dimension total score range from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better QoL. Overall score can be summarized in the Parkinson's Disease Summary Index (PDSI) or PDQ-39 Summary Index (PDQ-39 SI).PDSI or PDQ-39 SI = sum of dimension total scores divided by 8 which then reflects a mean score ranging from 0 to 19.5 with a lower number reflecting better quality of life.
Time Frame: Baseline and End of Study - 2 Months
Population: One participant was dropped from the analysis due to cognitive impairment and difficulty completing the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMPOWER PD Clinic Participation
Number analyzed (Participants) | 18
score on a scale
  PDQ-39 SI Pre Assess | 3.93 (2.27)
  PDQ-39 SI Post Assess | 4.22 (2.60)
Statistical Analysis 1: Comparison: EMPOWER PD Clinic Participation; Test type: Other; p = 0.309, t-test, 2 sided

9. Secondary Outcome: Change in the Parkinson's Fatigue Scale (PFS-16).
Description: The PFS-16 is a 16-item patient rated scale based on feelings and experiences over the past two weeks. Seven items tap the presence or absence of the subjective experience of fatigue with an emphasis on the physical effects of fatigue and nine items address the impact of fatigue on daily functioning and activities, including socialization and work but not exercise specifically. Scoring options range from 1 ("strongly disagree") to 5 (strongly agree"). A total ordinal PFS score ranging from 16-80 based on the sum of the scores will be used.
Time Frame: Baseline and End of Study - 2 Months
Population: One participant was dropped from the analysis due to cognitive impairment and difficulty completing the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMPOWER PD Clinic Participation
Number analyzed (Participants) | 18
score on a scale
  PFS-16 Pre Assess | 40.39 (14.01)
  PFS-16 Post Assess | 40.67 (14.39)
Statistical Analysis 1: Comparison: EMPOWER PD Clinic Participation; Test type: Other; p = 0.827, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 months
Description: Other adverse event would include events that occurred during the time participants were actively engaged in the clinic or educational intervention such as falls or any other reported medical event.
Arm/Group | EMPOWER PD Clinic Participation
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol: Study Protocol and Statistical Analysis Plan (2024-07-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT05640167/Prot_000.pdf
  • Study Protocol and Statistical Analysis Plan: Study Protocol and Statistical Analysis Plan Original (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT05640167/Prot_SAP_001.pdf